CLINICAL TRIAL: NCT04464681
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Continuous Intravenous Injection, Dose Escalation, Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of M201-A in Healthy Japanese Subjects
Brief Title: Multiple Dose Escalation Study of M201-A in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kitasato University (Other)
Collaborators: Aetas Pharma Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Tomoko Hasunuma, Director of Clinical Trial Center, Kitasato University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M201-A-CT-003
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M201-A Injection (Experimental): Active Substance: M201-A Route of administration: continuous intravenous injection
  Interventions: Drug: M201-A Injection
- Placebo (Placebo Comparator): Placebo: M201-A Placebo Route of administration: continuous intravenous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M201-A Injection — Active Substance: M201-A Route of administration: continuous intravenous injection
  Arms: M201-A Injection
Drug: Placebo — Placebo: M201-A Placebo Route of administration: continuous intravenous injection
  Arms: Placebo

SUMMARY:
This Phase I is designed to evaluate the safety, tolerability and pharmacokinetics of multiple ascending doses of M201-A administered by multiple continuous intravenous injection in Healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study

* (1)Japanese Healthy Male subjects
* (2)Age 20 to less than 50 years of age
* (3)Body Weight of more than 50 kg, Body Mass Index (BMI) of 18.5 to less than 25.0 kg/m2 at the screening examination
* (4)Written informed consent must be obtained on a voluntary basis before any assessment is performed.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

* (1)Presence or past medical history of hepatic impairments, renal impairments, cardiovascular disease, gastrointestinal disease and others which are inappropriate for participating in this clinical trial
* (2)Past medical history of cancer, cerebral infarction or cardiac infarction
* (3)Past history of surgical operation of gastrointestine or kidney except appendectomy or hemorrhoid operation.
* (4)Presence or past history of epilepsy.
* (5)Presence or past medical history of allergic reactions or idiosyncrasies to food, medicinal substance and metallic materials
* (6)heart rate(HR) >= 100 bpm at the screening examination
* (7)The corrected QT interval(QTcF) >= 440 ms at the screening examination
* (8)brain natriuretic peptide(BNP) > 40 pg/mL at the screening examination
* (9)K<3.6 mEq/L at the screening examination
* (10)Past history or suspect of aldosteronism.
* (11)Any risk factors of Torsades de Pointes including such as heart failure, hypokalemia, long QT interval syndrome due to family medical history
* (12)Cre>1.10 mg/dL, <0.85 mg/dL at the screening examination
* (13)Subject who donated whole blood of 400 mL within 12 weeks or whole blood of 400 mL of 200 mL / blood component donation within 4weeks prior to the first administration.
* (14)Use of prescription drug, over-the-counter medications (except eye drops for dryness, sanitizer for preventing infection), or herbal medication within 4 weeks prior to study medication.
* (15)Subject who consumed furanocoumarin containing food within 7 days prior to study medication.
* (16)Subject who drunk alcohol or caffeine containing drink within 3 days prior to study medication.
* (17)Subject who was administered of another investigational drug within16 weeks prior to agree to participate in this study.
* (18)Subject who was administered M201-A in the past.
* (19)Subject who smoke within 90 day prior to study medication or who cannot quit smoking during the study period.
* (20)Subject with positive result in hepatitis B(HB)s antigen, hepatitis C virus(HCV) antibody, HIV antigen/antibody, Syphilis serum, urine drug test at the screening test. Subject with positive result in Coronavirus(COVID-19) test at the screening or at the hospitalization.
* (21) Presence or past history of drug/alcohol abuse.
* (22)Subject who do not use medically acceptable contraceptive method until 90 days after the final study drug administration.
* (23)Subject who investigator judges ineligible for other reasons

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Throughout the study duration up to day 11
  Number of participants with adverse events, serious adverse events, physical examinations, vital sign measurements, 12-lead ECGs, Holter ECG, clinical laboratory safety tests (including hematology, chemistry, and urinalysis), recording of concomitant medications and procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Department of Research, KITASATO UNIVERSITY KITASATO INSTITUTE HOSPITAL, Tokyo, Japan